CLINICAL TRIAL: NCT03835806
Title: Blister Eradication Looking at Impact of Experimental Versus Established Regimens
Acronym: BELIEVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Patrick B Burns, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-49612
Record Dates: First submitted 2019-02-02; First posted 2019-02-11 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Blister of Foot

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial looking at a novel blister treatment intervention versus a traditional model.
Masking Description: The treatments are visually dissimilar, therefore blinding for the investigator and subject is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastikon - traditional (Active Comparator): The participant will be randomized to a treatment arm according to their racing bib number. Even bib numbers will be in the Elastikon treatment arm. The researcher will evaluate the blister and treat according to treatment arm with the following blister treatment device intervention: the blister will be prepped per routine, drained, covered with paper tape, sprayed with adhesive spray and then covered with Elastikon.
  Interventions: Other: Elastikon
- Rocktape - novel (Experimental): The participant will be randomized to a treatment arm according to their racing bib number. Odd bib numbers will be in the Rocktape treatment arm. The researcher will evaluate the blister and treat according to treatment arm with the following blister treatment device intervention: the blister will be prepped per routine, drained, covered with paper tape and then covered with Rocktape
  Interventions: Other: Rocktape

INTERVENTIONS:
Other: Elastikon — This randomized controlled trial will compare the traditional method of treating blisters with a multi-step approach of percutaneous drainage, paper tape, spray adhesive and then Elastikon which is our traditional blister treatment approach.
  Arms: Elastikon - traditional
Other: Rocktape — This randomized controlled trial will compare the traditional method of treating blisters with a multi-step approach of percutaneous drainage, paper tape and then Rocktape which is our novel blister treatment approach.
  Arms: Rocktape - novel

SUMMARY:
The specific aim of this study is to evaluate whether RockTape has similar efficacy to Elastikon in the treatment of foot blisters in ultramarathon runners. Elastikon with paper tape and spray adhesive is a well-accepted means of blister treatment and has been used by medical staff at over 50 multi-stage ultramarathons around the world. RockTape is another commercially available product that has also been used by runners successfully to treat foot blisters. RockTape's adhesive qualities have a potential advantage over Elastikon, in that it does not require an additional adhesive substituting a level of complexity, weight, and cost for foot care. There have been no studies examining the efficacy of either agent for blister treatment.

This randomized controlled trial will compare the traditional method of treating blisters with a multi-step approach of percutaneous drainage, paper tape, spray adhesive and then Elastikon to percutaneous drainage, paper tape and RockTape.

DETAILED DESCRIPTION:
Friction foot blisters are one of the most common injuries encountered by hikers and runners(1) with incidence as high as 39% in marathoners(2). In adventure races it is the most commonly reported injury(3) and in expedition length ultramarathons, blisters account for nearly 74% of medical visits(4). While most blisters are of minor medical significance, they can impair concentration, decrease athletic performance, and can be potentially debilitating.

The specific aim of this study is to evaluate whether RockTape has similar efficacy to Elastikon in the treatment of foot blisters in ultramarathon runners. Elastikon with paper tape and spray adhesive is a well-accepted means of blister treatment and has been used by medical staff at over 50 multi-stage ultramarathons around the world. RockTape is another commercially available product that has also been used by runners successfully to treat foot blisters. RockTape's adhesive qualities have a potential advantage over Elastikon, in that it does not require an additional adhesive substituting a level of complexity, weight, and cost for foot care. There have been no studies examining the efficacy of either agent for blister treatment.

This randomized controlled trial will compare the traditional method of treating blisters with a multi-step approach of percutaneous drainage, paper tape, spray adhesive and then Elastikon to percutaneous drainage, paper tape and RockTape.

ELIGIBILITY:
Inclusion Criteria:

* The study enrollment period will run for approximately 7 days over 3 weeks throughout 2019 at Racing the Planet races in Namibia, Mongolia and Chile. All racers are potential subjects.

Subjects will be enrolled when they present to the medical tent for the treatment of their first painful blister. The subject will be evaluated for exclusion criteria and the subject will be asked to select the most painful blister to be included in the study. All other blisters may be treated through traditional means and are not included in the study.

Exclusion Criteria:

* Blister exclusion criteria:

  1. Toe blisters will be excluded because they are treated with paper tape only to avoid friction against neighboring toes and further blister formation.
  2. Only intact blisters are included in this study as de-roofed blisters are treated differently.
  3. Hemorrhagic blisters are excluded as they are often not amenable to percutaneous drainage given the increased risk in infection.

If the most painful blister is a toe blister or a hemorrhagic blister, then the second most painful blister will be selected. If there is no second blister, the subject cannot be enrolled at this time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-04-27 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success | Data will be collected during the 1 week ultramarathon in austere conditions until study completion, usually 3-5 days. This will be conducted over 3 separate races.
  The subject's involvement in the study will end in one of the following situations and the researcher will fill out the appropriate data sheet at the time of the subject's departure from the study.
  1. The blister treatment is a success as defined by:
     1. the blister treatment falls off and the subject has no pain and no blister reoccurrence
     2. the blister treatment is removed by the subject and does not need to be replaced because the there is no pain or blister present
     3. the blister treatment stays on for the length of the study needing no intervention
  2. The blister treatment is a failure as defined by:
     1. if the blister re-occurs
     2. if the treated area has pain to the point that the blister treatment must be removed to evaluate
     3. if the subject removes the blister treatment and needs to be retreated.
  3. The race has come to completion
  4. The subject withdraws from the race or the study.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick B Burns, MD, Principal Investigator — Stanford University
Locations (3):
- Racing the Planet, San Pedro de Atacama, Chile
- Racing the Planet, Ulaanbaatar, Mongolia
- Namib Desert, Windhoek, Namibia

IPD SHARING:
Plan to Share IPD: No